CLINICAL TRIAL: NCT03609749
Title: Mindfulness Influences on Self-Regulation: Mindful Self-Regulation fMRI Study
Brief Title: Mindful Self-Regulation fMRI Study (MindfulPCfMRI)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Martinos Center for Biomedical Imaging (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH); Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHA-IRB-1002/08/14_fMRI; UH2AT009145 (NIH)
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Primary Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Training for Primary Care (Experimental): Experimental: Mindfulness Training for Primary Care For intervention description see Mindfulness Training for Primary Care (MTPC) in the study "MINDFUL-PC: Integrating Mindfulness Into the Patient-Centered Medical Home (Phase 3)". For the Mindfulness Training for Primary Care (MTPC) fMRI - arm, the investigators acquire pre-/post-intervention neuroimaging measures from subjects enrolled in this additional fMRI study.
  Interventions: Behavioral: Mindfulness Training for Primary Care

INTERVENTIONS:
Behavioral: Mindfulness Training for Primary Care — For intervention description see Mindfulness Training for Primary Care (MTPC) in the study "MINDFUL-PC: Integrating Mindfulness Into the Patient-Centered Medical Home (Phase 3)"

SUMMARY:
The purpose of this study is to investigate changes in functional neural activation during self-regulation tasks before compared to after the Mindfulness Training for Primary Care intervention (see MINDFUL-PC (Phase 3) clinical trial). The study will also look at whether chronic disease self-management action plan initiation and successful engagement of self-report and behavioral self-regulation targets relates to the observed brain activation changes after compared to before the mindfulness intervention.

DETAILED DESCRIPTION:
The investigators will investigate the effects of MTPC on pre/post changes in neural function with self-regulation target engagement, using self-appraisal, cuff pain and pain anticipation, and interoceptive attention fMRI tasks among primary care patients with an anxiety or depressive disorder. Primary outcome for this study is evaluating the changes in OFC activation during self-criticism blocks within a self-appraisal fMRI task. Secondary outcomes include changes in activation during self-appraisal fMRI task, pain regulation task, and interoceptive attention task, and the relationship of these targets with medical regimen adherence.

ELIGIBILITY:
Inclusion Criteria:

(In addition to all of the inclusion criteria for the main study, see MINDFUL-PC: Integrating Mindfulness into the Patient-Centered Medical Home (Phase 3))

1. Adults 21-60 years old enrolled for participation in the MINDFUL-PC study.
2. During baseline visit, patient has a history of either major depressive disorder, dysthymia, or generalized anxiety disorder, OR has current mild to moderate symptoms of depression (score range of 10-28 on DASS-21 Depression subscale) or anxiety (score >7 on DASS-21 anxiety subscale).
3. Does not have a substance use disorder nor intoxication at the time of scanning. Patients must report no more than infrequent recreational cannabis use (i.e., no more than two times a month) and must report capacity for abstinence from both cannabis and ethyl alcohol for the 72 hours prior to the scan.
4. Normal or corrected-to-normal vision, and correction must be with contact lenses.
5. Right-handed as defined by Edinburgh Handedness Inventory.

Exclusion Criteria:

1. Current severe panic disorder, active severe PTSD symptoms, or psychosis.
2. Current suicidality OR severe depression as evidenced by a score of 28 or higher on the DASS-21 Depression subscale.
3. Standard direct exclusion criteria for undergoing magnetic resonance imaging (MRI) procedures for research purposes (safety standards), i.e., Meniere's disease, epilepsy, strong claustrophobia, currently pregnant or breastfeeding or planning to conceive or breastfeed during the study, cardiac pacemaker, prosthetic heart valve, neurostimulator, implanted pumps, non-MR-compatible implants or devices.
4. A history of neurological disease or injury, including a history of seizures or significant head trauma (i.e., extended loss of consciousness, neurological sequelae, or known structural brain lesion), or previous brain surgery. These participants are excluded because they may confound the results of the study due to potential abnormalities in their nervous system.
5. Severe skin disease, skin allergies, or multiple reactions to topical preparations, dressings or tapes (because we will be placing sensors on the skin to record cardiac activity and skin conductance).
6. Age greater than 60 years old because age effects may confound the results of the study, because white matter integrity decreases with age and reduced inhibitory control.
7. Current meditation or intense yoga practice of more than 10 minutes a day of current mindfulness meditation practice, 200 hours of total lifetime meditation practice (non-MBI), or more than 63 lifetime hours of MBI-related mindfulness practice.
8. Participants with body weight >230 lbs or BMI > 38 will require additional in-person screening and PI approval, because of potential tight fit in the MRI scanner.
9. Participants with vascular disease, such as peripheral vascular disease, varicose veins, or lymphedema, in both lower limbs.
10. Based on clinical judgment and safety assessment by the PI, the participant is inappropriate for fMRI or unable to complete experiments.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Change in orbitofrontal cortex activation during the self-criticism condition in self-appraisal task | Weeks 8 - 10
  This task involves asking the participant to read about situations and imagine him/herself being self-critical or self-reassuring in these conditions.

SECONDARY OUTCOMES:
Change in insula activation during an interoceptive attention task | Weeks 8 - 10
  This task contrasts an interoceptive attention condition with an exteroceptive attention condition.
Changes in the rostral anterior cingulate cortex and adjacent medial prefrontal cortex (rACC/mPFC) during the anticipation of pain | Weeks 8 - 10
  This task involves a pressure cuff which is placed on participant's calf and is inflated for periods of 30 seconds to a medium intense pain, as rated by the participants.
Change in activation of the medial prefrontal cortex during the self-criticism condition in self-appraisal task | Weeks 8 - 10
  This task involves asking the participant to read about situations and imagine him/herself being self-critical or self-reassuring in these conditions.
Correlations between brain activation changes and chronic disease self-management action plan initiation | Weeks 8 - 10
  Patient self-reported Action Plan Initiation Survey (APIS-5) is a 5-item questionnaire in which patients are asked to list their action plan SMART goal created during the study, and determine whether they met or did not meet the goal using a 7-point Likert scale with scores >=5 representing self-reported initiation of the goal.

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance Center for Mindfulness and Compassion, Somerville, Massachusetts, United States

REFERENCES:
- [Background] Longe O, Maratos FA, Gilbert P, Evans G, Volker F, Rockliff H, Rippon G. Having a word with yourself: neural correlates of self-criticism and self-reassurance. Neuroimage. 2010 Jan 15;49(2):1849-56. doi: 10.1016/j.neuroimage.2009.09.019. Epub 2009 Sep 18. PMID 19770047
- [Background] Farb NA, Segal ZV, Anderson AK. Mindfulness meditation training alters cortical representations of interoceptive attention. Soc Cogn Affect Neurosci. 2013 Jan;8(1):15-26. doi: 10.1093/scan/nss066. Epub 2012 Jun 11. PMID 22689216
- [Background] Loggia ML, Berna C, Kim J, Cahalan CM, Gollub RL, Wasan AD, Harris RE, Edwards RR, Napadow V. Disrupted brain circuitry for pain-related reward/punishment in fibromyalgia. Arthritis Rheumatol. 2014 Jan;66(1):203-12. doi: 10.1002/art.38191. PMID 24449585

DOCUMENTS (1):
  • Informed Consent Form (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT03609749/ICF_000.pdf